CLINICAL TRIAL: NCT06825221
Title: Novel Immune-modulating Formula Versus Standard Formula for Malnourished Gastrointestinal Cancer Patients Undergoing Cancer Surgery: A Randomized Controlled Trial.
Brief Title: Effect of Immune Formula in Gastrointestinal Cancer Patients Undergoing Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0711/65
Record Dates: First submitted 2025-02-10; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Malnutrition; Cancer
MeSH Terms: conditions — Malnutrition; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: * The same sachet, taste, and appearance for both formula
  * Care provider and outcome assessor will be blinded for study arm of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants receive 2 packages of immune formula per day for 10-14 days + dietary counseling
  Interventions: Dietary Supplement: Oral Nutrition supplement
- Control group (No Intervention): Participants receive 2 packages of standard formula per day for 10-14 days + dietary counseling

INTERVENTIONS:
Dietary Supplement: Oral Nutrition supplement — Participants received normal diet and in the interventional group received package of immune formula 2 meals per day for 10-14 days prior surgery.
  Other Names: Immune formula
  Arms: Intervention group

SUMMARY:
Malnutrition is a common feature in cancer patients and associated with worse outcomes especially increased risk of postoperative complications in patients undergoing surgery.

The European Society for Clinical Nutrition and Metabolism (ESPEN) recommends preoperative oral/enteral immunonutrition support to decrease risk of postoperative complications. However, the evidence comparing between immune formula and standard formula is still controversial. Numerous studies have indicated that curcumin is beneficial to the immune system. This study aimed to assess the effect of an immune formula which contains curcumin versus standard formula for malnourished gastrointestinal cancer patients undergoing cancer surgery.

A randomized controlled trial will be conducted on 40 malnourished gastrointestinal cancer patients who plan to undergo major cancer surgery. Patients in the intervention group will receive 2 sachets of immune formula per day (355.5 kcal and curcumin 25 mg per sachet) for 10-14 days and dietary counseling. Participants in the control group will receive 2 sachets of isocaloric standard formula per day for 10-14 days and dietary counseling. Anthropometry and biochemical parameters were measured in 3 periods (before intervention, two weeks after intervention in preoperative, and post-operative period). Postoperative complications were recorded until patient discharge from hospital for 30 days.

DETAILED DESCRIPTION:
Malnutrition is a common feature in cancer patients and associated with worse outcomes especially increased risk of postoperative complications in patients undergoing surgery.

The European Society for Clinical Nutrition and Metabolism (ESPEN) recommends preoperative oral/enteral immunonutrition support to decrease risk of postoperative complications especially in malnourished patients undergoing major abdominal surgery. Numerous studies have indicated that curcumin is beneficial to the immune system. This study aimed to assess the effect of an immune formula which contains curcumin versus standard formula for malnourished gastrointestinal cancer patients undergoing cancer surgery.

A randomized controlled trial will be conducted on 40 malnourished gastrointestinal cancer patients who plan to undergo major cancer surgery. Patients in the intervention group will receive 2 sachets of immune formula per day (355.5 kcal and curcumin 25 mg per sachet) for 10-14 days and dietary counseling. Participants in the control group will receive 2 sachets of isocaloric standard formula per day for 10-14 days and dietary counseling.

Body mass index (BMI), body composition, mid-arm muscle circumference (MAMC), hand grip strength, food intake, pre-albumin, C-reactive protein (CRP), Interleukin-6 (IL-6), and Tumor necrosis factor alpha (TNF-alpha) are measured at the day before and the day after having all of oral nutrition supplements. Parameters are re-measured within 5-7 days after operation along with fasting blood sugar, insulin and HOMAR-IR. Postoperative complications are assessed with Clavien-Dindo classification on the last day in the hospital. Re-admit rates are recorded until 30 days after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Participants who were malnourished gastrointestinal cancer patients and plan to treatment with surgery
* Participant aged ≥18 years

Exclusion Criteria:

* Participants who weren't willing to participate in a clinical trial.
* Participants who were pregnant or lactating
* Participants who were enteral feeding intolerance such as gastrointestinal obstruction
* Participants who receive jejunal feeding
* Participant has been taking an immune formula prior to the baseline visit.
* Participants who were allergic to components of the study formula such as milk,soy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change in C-reactive protein | Baseline,Study day 10-14, After surgery day 5-7
  C-reactive protein in mg/L
Change in Tumor necrosis factor alpha (TNF-α) | Baseline,Study day 10-14, After surgery day 5-7
  Tumor necrosis factor alpha in pg/ml
Change in interleukin-6 (IL-6) | Baseline,Study day 10-14, After surgery day 5-7
  Interleukin-6 in pg/ml

SECONDARY OUTCOMES:
Change in Prealbumin | Baseline,Study day 10-14, After surgery day 5-7
  Prealbumin in (g/L)
Mid-upper arm circumference | Baseline,Study day 10-14, After surgery day 5-7
  MAMC in cm
BIA | Baseline,Study day 10-14, After surgery day 5-7
  BIA is body composition analysis in muscle mass, fat mass,% body fat
Handgrip strength | Baseline,Study day 10-14, After surgery day 5-7
  Handgrip strength in kg
Complication during hospitalized stay | Hospital stay
  Complication assessment by Clavien-Dindo classification
Rate of death during hospitalized stay | Hospital stay
  Check number of participants at death during hospitalized stay
Rate of re-admission within 30 days | 30 day after discharge
  Check re-admission within 30 days after discharge
Fasting blood glucose | After surgery day 5-7
  Fasting blood glucose in mg/dL
Insulin (Homa IR) | After surgery day 5-7
Gastrointestinal tolerance | Baseline,Study day 10-14
  Gastrointestinal tolerance including abdominal distention,nausea,vomiting and diarrhea

CONTACTS AND LOCATIONS:
Overall Officials: Narisorn Lakananurak, Doctor, Principal Investigator — Chulalongkorn University
Locations (1):
- Department of Medicine, Chulalongkorn University, Bangkok, Thailand

REFERENCES:
- [Derived] Lakananurak N, Laosuwan P, Vongwattanakit P, Jittivasurat A, Techasukthavorn V. Novel Immune-Modulating Formula Versus Standard Formula for Gastrointestinal Cancer Patients at Risk of Malnutrition Undergoing Surgery: A Pilot Randomized Controlled Trial. Clin Nutr ESPEN. 2026 Jan 10:102909. doi: 10.1016/j.clnesp.2026.102909. Online ahead of print. PMID 41525872